CLINICAL TRIAL: NCT01314885
Title: Randomized, Double-Blind, Double-Dummy, Placebo-Controlled, 3-Way Crossover Study To Determine The Effects Of Single Inhaled Doses Of PF-03715455 (20 Mg) And PH-797804 (30 Mg) On Induced Sputum Neutrophils Following Inhaled Lipopolysaccharide (LPS) Challenge In Healthy Volunteers
Brief Title: Single Dose Lipopolysaccharide (LPS) Study In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: A9111003
Record Dates: First submitted 2010-11-05; First posted 2011-03-15 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Healthy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — N-(1-(3-chloro-4-hydroxyphenyl)-3-(1,1-dimethylethyl)-1H-pyrazol-5-yl)-N'-((2-((3-(2-((2-hydroxyethyl)thio)phenyl)-1,2,4-triazolo(4,3-a)pyridin-6-yl)thio)phenyl)methyl)-urea; PH 797804

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-03715455 (Experimental)
  Interventions: Drug: PF-03715455
- PH-797804 (Experimental)
  Interventions: Drug: PH-797804
- Placebo for PF-03715455 (Placebo Comparator)
  Interventions: Drug: Placebo for PF-03715455
- Placebo for PH-797804 (Placebo Comparator)
  Interventions: Drug: Placebo for PH-797804

INTERVENTIONS:
Drug: PF-03715455 — 20mg, Inhaled, single dose
  Arms: PF-03715455
Drug: PH-797804 — 30mg, Oral, single dose
  Arms: PH-797804
Drug: Placebo for PF-03715455 — Single dose, inhaled, Placebo for PF-03715455
  Arms: Placebo for PF-03715455
Drug: Placebo for PH-797804 — Single Dose, Oral, Placebo for PH-797804
  Arms: Placebo for PH-797804

SUMMARY:
A single dose study with the inhaled anti-inflammatory agent PF-03715455 to establish if it has anti-inflammatory activity following a challenge with LPS. Inhaled LPS invokes an acute inflammatory response in the lung which can be seen in induced sputum. PH-0797804 is an internal control for the study.

DETAILED DESCRIPTION:
Proof of Mechanism

ELIGIBILITY:
Inclusion Criteria:

* Male or female (of non-child bearing potential) subjects, aged 18-50 years.
* Subjects whose FEV1 and FVC at screening are both greater than or equal to 80% of their predicted value for age, race, sex and height.
* Subjects who have normoresponsive airways.
* Subjects who are able to successfully complete screening sputum inductions.

Exclusion Criteria:

* Subjects who have evidence, on review of pre-study laboratory data and full physical examination, or history of any clinically significant hematological, renal, endocrine, gastrointestinal, dermatological, hepatic, psychiatric, neurologic diseases. Specifically liver function tests and CRP must be within the reference range.
* Subjects with a medical history of asthma symptomatology (ie, wheeze and/or dyspnea at rest).
* Subjects who have experienced a respiratory tract infection within the previous 4 weeks or any other infection within 1 week of dosing

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Post LPS sputum neutrophil % is being evaluated at the end of each treatment period to establish the effect of treatment on this endpoint | 6 hours

SECONDARY OUTCOMES:
Cell counts, IL-6, MPO, MCP-1, MIP1b are individual endpoints which will be evaluated in sputum however they are collected as a single sample. | 6 hours
Post-LPS systemic inflammatory indices: Neutrophil count, IL-6, IL-10, MPO, MCP-1, MIP1b, fibrinogen, CC16 and CRP. These are individual endpoints which will be evaluated in blood however they are collected as a single sample. | 1, 4, 6 and 7 hours
Number of participants with adverse events | Baseline, Day 1 and Day 2
Change from baseline in ECG parameters | Baseline, Day 1 and Day 2
Change from baseline in BP parameters | Baseline, Day 1 and Day 2
Change from baseline in lab safety parameters | Baseline, Day 1 and Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United Kingdom (2):
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9111003&StudyName=Single%20Dose%20Lipopolysaccharide%20%28LPS%29%20Study%20In%20Healthy%20Volunteers